CLINICAL TRIAL: NCT06030284
Title: The True Efficacy of Burst Spinal Cord Stimulation in the Management of Intractable Low Back Pain
Brief Title: The True Efficacy of Burst Spinal Cord Stimulation in the Management of Intractable Low Back Pain (TRU-BURST)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision was taken to consider other opportunities for collecting sham-controlled data for BurstDR SCS.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABT-CIP-10453
Record Dates: First submitted 2023-08-11; First posted 2023-09-08 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-08

CONDITIONS: Chronic Intractable Pain
Keywords: ABT-CIP-10453; Spinal Cord Stimulation; TRU-BURST; BurstDR-SCS; FBSS

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BurstDR-SCS (Experimental): Subjects implanted with BurstDR-SCS will be included in BurstDR-SCS arm.
  Interventions: Device: BurstDR-SCS
- Sham control arm (Experimental): Subjects implanted with the BurstDR-SCS system will be included in the Sham control arm
  Interventions: Device: BurstDR-SCS

INTERVENTIONS:
Device: BurstDR-SCS — Spinal Cord Stimulation with a BurstDR-SCS system.
  Arms: BurstDR-SCS
Device: BurstDR-SCS — BurstDR-SCS system turned off.
  Arms: Sham control arm

SUMMARY:
The purpose of this prospective, multi-center, randomized, triple-blind, sham-controlled study with parallel economic evaluation is to test the analgesic superiority of BurstDR-SCS compared to sham stimulation using both traditional patient-reported pain outcome measures and objective physiologic data collected from patient-worn biosensors. The endpoints associated with these objectives will be studied across a follow-up period of 6 months.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation-related procedure.
2. Subject is at least 18 years of age or older at the time of enrollment.
3. Subject is a potential candidate for trial of an Abbott neuromodulation SCS system for chronic intractable pain and is able to engage in the use of wearables and surveys at least 9 days before commencing their neuromodulation trial period.
4. Subject is willing to undergo a temporary trial of the Abbott neuromodulation SCS system lasting at least 7 days.
5. Subject's average low back pain intensity is ≥ 6 out of 10 on pain numerical rating scale (NRS).
6. Subject has Failed Back Surgery Syndrome (FBSS with persistent low back pain for ≥ 6 months following lumbar spine surgery). OR Subject has not had spine or back surgery AND subject has chronic (at least 6 months), refractory axial low back pain with a neuropathic component, AND subject is not a candidate for spine surgery (recommended to have an orthopedic surgeon review patient's imaging and confirm this).
7. Subject's leg pain NRS, if present, is less than or equal to back pain NRS.
8. Subject is on stable pain medications, as determined by the Investigator, for at least 28 days prior to enrolling in this study and agrees to not change medication dosage without consulting Investigator.
9. Subject agrees not to introduce or change other therapies related to pain without consulting investigator (e.g., physical therapy, psychotherapy, medical interventions). Rescue analgesic medication for chronic pain or for non-index pain (e.g., ibuprofen for an ankle sprain) will be allowed but must be reported.
10. Subject agrees to report on any healthcare received during the study period.
11. Subject is willing to cooperate with all study requirements including completion of office visits, use of the wearable biosensors during daily activities, regular response to electronic surveys via the iPhone, and use of an at-home medication tracking log for tracking analgesic use and at-home healthcare tracking log (according to schedule outlined in section 6.0 of the protocol).
12. Subject understands that if they are enrolled, they will receive SCS during the trial period before receiving permanent implant. If they continue to a permanent implant, they will be randomly assigned to either sham stimulation or normal stimulation (50% chance) for a period of 6 months.
13. Subject understands that at study completion the implanted SCS system will not be explanted or removed as part of the study, regardless of study outcomes.

General Exclusion Criteria:

1. Subject is not willing to receive implant of a primary cell SCS system.
2. Subject is taking more than 50 morphine equivalents of opioid per day.
3. Subject has an unstable fusion with FBSS.
4. Subject's back and/or leg pain is believed to originate from spinal instability/mechanical pain.
5. Subject's back and/or leg pain is believed to originate from existing metal work.
6. Subject's low back pain is limited to a single focal pain area that suggests mechanical back pain.
7. Subject is currently participating, or intends to participate in another clinical investigation investigating pain management or that could present a confound to this study (per the investigator).
8. Subject is pregnant or nursing or subject plans pregnancy during the clinical investigation follow-up period. This includes female who is sexually active and not using a reliable form of birth control or being not surgically sterile or subject is listed as a post-menopausal female within less than 1 year.
9. Subject is part of a vulnerable population ( as per section 5.2.2.1 of the study protocol).
10. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation.
11. Subject has chronic widespread pain or confounding pain that will interfere with reporting of low back and leg pain (e.g. consider any chronic pain in the upper back, neck, head, face, shoulders, arms, or chronic headaches)
12. Subject has previously had permanent implantation of another SCS, DRG stimulation, or intrathecal drug delivery system or is scheduled to receive such system in a timeframe that would overlap with this study.
13. Subject has already participated in a SCS trial period before enrolling in the study and is now waiting for their permanent implantation.
14. Subject engages in a profession or other activity that could be damaging to the wearable sensors, as determined by the investigator.
15. Subject has a skin condition that could be exacerbated by use of the wearable biosensors (e.g., skin allergy to metals, plastics), as determined by the investigator.
16. Subject has a physical condition that makes it difficult to wear the wearable sensors, as determined by the investigator.
17. Subject is bedridden.
18. Subject has life expectancy of less than 12 months.
19. Subject has a current diagnosis of a progressive neurological disorder as determined by the investigator. (e.g. multiple sclerosis, Huntington's disease)
20. Subject has a bleeding diathesis such as coagulopathy or thrombocytopenia
21. Subject has a current diagnosis of a coagulation disorder or uncontrolled diabetes mellitus.
22. Subject is immunocompromised and at an increased risk for infection
23. Subject has a systemic infection or local infection
24. Subject has regular intake of systemic steroids (except inhaled steroids used to treat asthma)
25. BMI > 40.
26. Subject has an active malignant disease or history of cancer requiring treatment in the last 12 months.
27. Evidence of an active disruptive psychological or psychiatric disorder or social condition as determined by the investigator.
28. Suspicion or evidence of untreated mental illness, substance abuse, or drug-seeking behavior.
29. Subject is involved in an injury claim under active litigation that involves back or leg pain/injury or is receiving or planning to receive worker's compensation payments related to back or leg pain.
30. Subject has a diagnosis of spondylolisthesis or scoliosis

Protocol-Specific Screening Exclusion Criteria:

1. Urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in overall back pain severity (NRS) at 6 months compared to sham arm | At 6 Months
  The pain severity endpoint is based on a review of previous RCTs of SCS and a consideration of IMMPACT (Initiative on Methods, Measurement and Pain Assessment in Clinical Trials) and COMET recommendations
Change in a composite of physiologic and behavioral features compared to sham arm leading up to 6 months post-permanent implant | At 6 Months
  Ability to use composite of physiologic and behavioral features (including data from biosensors) to identify treatment responders and physiological data collected from patient-worn biosensors.

SECONDARY OUTCOMES:
Change in percentage of patients reporting 50% or more reduction in backpain severity (NRS) at 6 months in treatment vs. sham | At 6 Months
Change in cumulative proportion of responders for back pain (NRS) in treatment vs. sham | At 6 Months
Change in pain-related catastrophizing (Pain Catastrophizing Scale) in treatment vs. sham | At 6 Months
  The Pain Catastrophizing Scale questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The questionnaire includes thirteen statements describing different thoughts and feelings that may be associated with pain. Using the scale 0-4 (0- not at all; 1- to a slight degree; 2- to a moderate degree; 3- to a great degree; and 4- all the time), the patients are expected to indicate the degree to which they have these thoughts and feelings when they're experiencing pain.
Change in functional disability (Oswestry Disability Index) in treatment vs. sham | At 6 Months
  The Oswestry Disability Index questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. An interpretation of 0% to 20% means minimal disability; 21% to 40% means moderate disability; 41% to 60% means severe disability; 61% to 80% means crippled; and 81%-100% means bed-bound patients.
Change in patient satisfaction (Patient Global Impression of Change) in treatment vs. sham | At 6 Months
  The Patient Global Impression of Change questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The scale ranges include:
  1. No change (or condition has gotten worse)
  2. Almost the same, hardly any change at all
  3. A little better, but no noticeable change
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better, and a slight but noticeable change
  6. Better and a definite improvement that has made a real and worthwhile difference
  7. A great deal better and a considerable improvement that has made all the difference
Change in health-related quality of life (EQ5D-5L) in treatment vs. sham | At 6 Months
  The EQ5D-5L questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints and to estimate health-related quality of life and quality-adjusted life years. It is a 5-level version of the EQ5D. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Change in health-related quality of life (PROMIS-29+2) in treatment vs. sham | At 6 Months
  The PROMIS-29+2 questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Change in emotional functioning improvement (Patient Health Questionnaire-9) in treatment vs. sham | At 6 Months
  The Patient Health Questionnaire-9 will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The Patient Health Questionnaire is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. It is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Change in pain interference PROMIS-29+2 domain in treatment vs. sham | At 6 Months
  The PROMIS-29+2 questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Change in social roles and activities PROMIS-29+2 domain in treatment vs. sham | At 6 Months
  The PROMIS-29+2 questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Change in sleep disturbance PROMIS-29+2 domain in treatment vs. sham | At 6 Months
  The PROMIS-29+2 questionnaire will be completed during selected clinical site visits via the electronic data acquisition portal. These questionnaires will be used for the assessment of study endpoints. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Change in on concomitant pain-related medication usage in treatment vs. sham | At 6 Months
  Importance of keeping pain-related treatments stable (per agreement with physician), including medications, physical therapy, psychotherapy, pain-related treatments (invasive or non-invasive) and interventions.
Change in overall leg pain severity (NRS) at 6 months compared to sham arm in patients who reported baseline chronic leg pain | At 6 Months
Change in percentage of patients reporting 50% or more reduction in leg pain severity (NRS) at 6 months in treatment vs. sham in patients who reported baseline chronic leg pain | At 6 Months
Change in cumulative proportion of responders for leg pain (NRS) in treatment vs. sham in patients who reported baseline chronic leg pain | At 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stefano Palmisani, Principal Investigator
Locations (5):
- Comprehensive Integrated Pain Program - Interventional Pain Service (CIPP-IPS) (Toronto Western Hospital), Toronto, Canada
- United Kingdom (4):
  - Seacroft Hospital, Leeds
  - The Walton Centre, Liverpool
  - Guy's and St. Thomas Hospital, London
  - St. Bartholomew Hospital, London

IPD SHARING:
Plan to Share IPD: No